CLINICAL TRIAL: NCT07380737
Title: Feasibility and Preliminary Effects of the Walking Tall App for Home-Based Gait Training in Parkinson's Disease: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0481_25_TLV_TG
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease
Keywords: Gait; Parkinson's Disease; Walking App; Rhythmic auditory cueing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Interventional Model: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walking Tall App Intervention (Experimental): Participants will use the Walking Tall smartphone app to complete 4-5 home-based walking sessions per week for 6 weeks. The app provides rhythmic auditory cues and verbal prompts to improve gait quality.
  Interventions: Behavioral: Walking Tall App

INTERVENTIONS:
Behavioral: Walking Tall App — Participants will use the Walking Tall smartphone app to complete 4-5 home-based walking sessions per week for 6 weeks. The app provides rhythmic auditory cues and verbal prompts to improve gait quality.

SUMMARY:
This is a pilot study designed to assess the feasibility, adherence, and preliminary effects of a 6-week home-based gait training intervention using the Walking Tall mobile app in individuals with Parkinson's disease. The app delivers rhythmic auditory cues and motivational verbal prompts to promote gait improvements. Primary outcomes include daily walking duration and step count measured via wearable sensors; secondary outcomes include gait speed, balance, self-reported confidence, and usability.

DETAILED DESCRIPTION:
This open-label, single-arm feasibility study will recruit 30 participants with idiopathic Parkinson's disease, currently enrolled in a rehabilitation program at the Ezra LeMarpe Organization in Israel. Participants will perform 4-5 walking sessions per week for 6 weeks using the Walking Tall smartphone application. The app delivers rhythmic cueing and motivational prompts to enhance walking speed, stride length, and confidence. The study includes baseline and post-intervention assessments. Walking behavior will be monitored using a tri-axial accelerometer worn for 7 days at each timepoint. The primary aim is to evaluate feasibility, adherence, and changes in daily walking activity, with secondary outcomes addressing gait parameters and user satisfaction. Findings will guide the design of future randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of idiopathic Parkinson's disease (MDS criteria)

Hoehn & Yahr stage II-III (ON-medication state)

Able to walk independently for ≥5 minutes

Stable medication for ≥1 month

Currently enrolled in a rehab program at Ezra LeMarpe

Able to provide written informed consent

Exclusion Criteria:

Musculoskeletal, neurological, or visual/hearing impairments affecting gait

Cognitive impairments or severe behavioral symptoms

History of stroke, severe TBI, or brain tumor

Cardiovascular contraindications

Inability to use a smartphone

Participation in other concurrent intervention studies

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Average Step Count Per Day | Time Frame: Baseline and 6 weeks
  Measured via accelerometer
Daily Walking Duration (minutes/week) | Time Frame: Baseline and 6 weeks
  Measured using tri-axial accelerometer (Axivity) over 7 days

SECONDARY OUTCOMES:
Gait Speed (m/s) - single- and dual-task | Time Frame: Baseline and 6 weeks
  Assessed using a 1-minute walking test under two conditions: (1) single-task (normal walking) and (2) dual-task (walking while performing a cognitive task such as serial subtraction). Gait speed is calculated in meters per second based on distance walked over time in each condition.
Short Physical Performance Battery (SPPB) | Time Frame: Baseline and 6 weeks
  The SPPB is a standardized test that evaluates lower extremity function using three components: balance (side-by-side, semi-tandem, tandem stance), gait speed over a 4-meter walk, and chair stands. Each component is scored from 0 to 4, with a total score ranging from 0 (worst performance) to 12 (best performance).
Timed Up and Go (TUG) - single- and dual-task | Time Frame: Baseline and 6 weeks
  The TUG test measures functional mobility by timing how long it takes a participant to stand up from a chair, walk 3 meters, turn, return, and sit down. It is performed under two conditions: (1) single-task (normal walking) and (2) dual-task (walking while performing a cognitive task, such as serial subtraction). The test evaluates gait, balance, and cognitive-motor integration.

OTHER OUTCOMES:
Self-reported questionnaires: Activities-specific Balance Confidence (ABC) | Time Frame: Baseline and 6 weeks
  Activities-specific Balance Confidence (ABC) Scale A 16-item self-report questionnaire assessing participants' confidence in performing various daily activities without losing balance or becoming unsteady. Scores range from 0% (no confidence) to 100% (complete confidence), with higher scores indicating greater balance confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Tatyana Gurevich, Prof, Principal Investigator — Head of the Movement Disorders Unit at Ichilov Hospital
Locations (1):
- Tel Aviv Sourasky Medical Center (Ichilov Hospital), Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brodie, M. A., & University of New South Wales. (2023, August 7). New app is a step towards helping people with Parkinson's disease walk more confidently. UNSW Newsroom. Retrieved from https://www.unsw.edu.au/newsroom/news/2023/08/new-app-is-a-step-towards-helping-people-with-parkinsons-disease